CLINICAL TRIAL: NCT06223867
Title: Evaluation of Efficacy, Effectiveness, and Implementation of Jaspr Health's Digital Platform in Emergency Department for Patients with Suicidal Risk- Part A: Randomized Controlled Trial
Brief Title: Efficacy, Effectiveness, and Implementation of Jaspr Health in Emergency Department- Part a
Acronym: Jaspr-PartA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Ohio State University (Other); Evidence-Based Practice Institute, Seattle, WA (Industry); Worcester Polytechnic Institute (Other); National Institute of Mental Health (NIMH) (NIH); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Edwin Boudreaux, Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00000716 Part A; 1P50MH129701 (NIH)
Record Dates: First submitted 2023-12-14; First posted 2024-01-25 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Suicidal Ideation; Suicide Attempt; Self Harm
Keywords: Suicide; Self-Harm; Attempt; Ideation; Suicidal thought; Suicidal plan; Crisis intervention; Suicide prevention; Emotional support; Mental Health; Behavioral Health; Psychiatry; Emergency Department; Technology; Mobile Application; Implementation; Safety Plan; Lethal Means
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted; Self-Injurious Behavior; Suicide; Suicide Prevention; Psychological Well-Being; Emergencies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome evaluators will be blinded to study condition. It is not possible to blind participants, the research staff enrolling the participant, or the treating clinicians.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Enhanced treatment as usual (ETAU) alone (Active Comparator): Subjects in this arm will receive the usual care for patients with suicidal risk at UMass Memorial ED that may include a behavioral health evaluation by a trained clinician, and environmental safety precautions dictated by risk level (Mild, Moderate, High). Individuals deemed appropriate for discharge undergo discharge planning and offered a personalized safety plan using the Stanley-Brown Safety Planning Intervention, including lethal means safety counseling.
  Interventions: Behavioral: ETAU
- Jaspr intervention with enhanced treatment as usual (ETAU) (Experimental): Subjects in this arm will receive ETAU in addition, they will complete a guided Suicide Status Interview (SSI), Safety Planning, and Lethal means counseling on the Jaspr tablet-based app before open access to the Jaspr resource library.
  Subjects can sign up to receive JAH mobile app.
  Interventions: Device: Jaspr App + JAH; Behavioral: ETAU

INTERVENTIONS:
Device: Jaspr App + JAH — With assistance form a research coordinator, the subject will complete self-administered suicide risk assessment on the tablet via Jaspr app, then the subject will engage with suicide-related coping skills and resources that the app provides. Subject will continue to have access to the coping skills and videos via a mobile app after discharge.
  Arms: Jaspr intervention with enhanced treatment as usual (ETAU)
Behavioral: ETAU — Usual care for suicidal patients at UMass Memorial ED that may include Behavioral health evaluation by a trained clinician. Environmental safety precautions. Personalized safety upon discharge
  Other Names: Enhanced Treatment As Usual

SUMMARY:
This Study will comprehensively evaluate a multi-component suicide prevention technology (Jaspr Health) that facilitates delivery of suicided-related evidence-based practices (EBPs) while replacing wasted waiting time with productive time in the Emergency Departments (EDs). The EBPs satisfy several key performance elements for systems adopting Zero Suicide.

A Complementary Randomized Controlled Trial and Real-World Study for Efficacy, Effectiveness, and Implementation Study Design (CREID) will be used

DETAILED DESCRIPTION:
This study will evaluate Jaspr's patient-facing tablet-based application (app) during suicide-related ED visits. The app guides patients in completing the Suicide Status Interview, which comprise of an evidence-based Collaborative Assessment & Management of Suicidality (CAMS) certified suicide prevention tools such as a suicide risk assessment, Stanley Brown- inspired safety planning, and lethal means safety counseling. It also offers access to a menu of "Comfort and Skills" modules that teaches patients behavioral skills to effectively manage imminent distress, while shared stories offer a library of professionally produced, racially and culturally diverse, inspirational videos of people with suicide-centered lived experience.

Subjects who interact with Jaspr can continue to access their safety plan, comfort and coping skills exercises, and the video library via Jaspr at Home (JAH) mobile application; a summary of the self-administered risk assessment is shared with the clinical team directly through the patient electronic medical record to help guide the treatment plan.

Part A of the study will be an individual, patient-level Randomized Controlled Trial (RCT) to evaluate the efficacy and mechanism of action of Jaspr's app intervention in EDs. All subjects will complete a baseline assessment prior to random assignment to one of the the two study conditions. All subjects will receive follow-up phone calls for 12 months after enrollment at weeks 6, 12, 24, 36, and 52. These calls will assess suicide related outcomes and healthcare utilization. In addition, the Massachusetts Department of Public Health (MA DPH) death registry will be reviewed, and each subject's electronic health record will be reviewed.

Part B of the study will be a Real-World Study (RWS) to evaluate the effectiveness and implementation processes in EDs and outcomes.

This ClinicalTrials.gov record will cover only Part A. Part B is summarized in a separate entry.

ELIGIBILITY:
Inclusion Criteria:

* Positive for suicide risk on the Patient Safety Screener in the ED (active suicidal ideation int the past 2 weeks, or suicidal attempt in the past 6 months)
* Cognitively and emotionally capable of consent and engaging in Jaspr app.
* Reads English at 6th grade level.
* Reliable telephone access.
* Owns a smart phone
* Lives in Massachusetts

Exclusion Criteria:

* Prisoners or in state custody
* Adults unable to consent
* Patient <18 yeas
* Enrolled subjects during the 12 month follow-up period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 670 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Suicide composite, binary | 12 months after enrollment
  Death by suicide OR suicide-related acute care utilization within 12 months after enrollment

SECONDARY OUTCOMES:
Suicidal attempt | 12 months after enrollment
  Suicidal attempt measured by the Columbia-Suicide Severity Rating Scale (CSSRS), Suicide attempt present Y/N
Suicidal behavior | 12 months after enrollment
  Suicidal behavior measured by the Columbia-Suicide Severity Rating Scale (CSSRS), including any preparatory, aborted, interrupted, and actual suicidal attempts. Suicidal Behavior present Y/N
Suicidal ideation severity | 12 months after enrollment
  Suicidal ideation severity measured by the Columbia-Suicide Severity Rating Scale (CSSRS). Suicidal Ideation (Highest Level Endorsed 1-5. 1= least severe and 5= highest severity)

OTHER OUTCOMES:
Evidence-Based Practice (EBP) delivery | During index visit= Day 1
  Number of patients receiving evidence based care, including evidence based suicide risk assessment, safety planning, lethal means safety counseling, cognitive behavioral therapy (CBT) coping skills training, suicide education materials, and behavioral health referral resources. Higher count = more EBPs delivered
Patient target engagement, perceived social support | 12 months after enrollment
  Perceived social support (attachment/affiliation) measured by Interpersonal Needs Questionnaire (INQ-15), Likert-type scale, higher scores = stronger social support
Patient target engagement, suicide-related coping | 12 months after enrollment
  Suicide-related coping (behavioral inhibition) measured by Suicide-Related Coping Scale (SRCS), Likert-type scale, higher scores = better ability to cope with suicidal thoughts
Patient target engagement, behavioral activation | 12 months after enrollment
  Behavioral activation (effort) measured by Behavioral Activation Scale (BAS) - Drive sub scale, Likert-type scale, higher scores = greater behavioral activation
In situ self-injury | Index visit= Day 1
  Intentional Self-Harm behavior during the index ED visit and inpatient stay related to the index visit, binary, In situ self-injury Yes/No
In situ distress | Index visit= Day 1
  Pre-post distress measure that will use 0 to 10 distress scale at start of enrollment and at 1, 2, 3 hours later. It will assess patient's distress during the index ED
In situ suicide related coping | Index visit= Day 1
  Pre-post suicide coping measure that will use 0 to 10 coping scale at start of enrollment and at 1, 2, 3 hours later. It will assess patient's suicide-related coping during the index ED
ED visit satisfaction | Index visit= Day 1
  0 to 10 visit satisfaction scale at start of enrollment and at 1, 2, 3 hours later to assess patient's satisfaction with the ED care during index visit
Psychiatric symptoms | Index visit and 12 months after enrollment
  Psychiatric symptoms on the diagnostic and statistical manual of mental disorders (DSM-5) Crosscutting measure, Likert-type scale, higher scores = more severe psychiatric symptoms
Patient reach | Duration of enrollment = 30 months
  Percentage of eligible patients who initiated Jaspr by answering at least one question on the Suicide Status Interview (SSI) in Jaspr app
Fidelity | Duration of enrollment = 30 months
  Percentage of patients who started the Suicide Status Interview (SSI) in Jaspr app and who completed the SSI and a safety plan (fidelity)
Exposure, time | Duration of enrollment = 30 months
  Within patients who started the Suicide Status Interview (SSI) in Jaspr app, total time spent on all components. Measured in minutes
Exposure, modules | Duration of enrollment = 30 months
  Within patients who started the Suicide Status Interview (SSI) in Jaspr app, total number of modules completed
Costs | Duration of enrollment = 30 months
  Costs associated with Jaspr preparation, training, deployment, use, workflow changes
Clinician acceptability | Duration of enrollment = 30 months
  Structured measure viewing Jaspr as agreeable, palatable, satisfactory using the Acceptability of Intervention Measure (AIM), Likert type scale, higher scores = stronger clinician acceptability
Patient acceptability | Duration of enrollment = 30 months
  Structured measure viewing Jaspr as agreeable, palatable, satisfactory using the Acceptability of Intervention Measure (AIM), Likert type scale, higher scores = stronger patient acceptability
Patient appropriateness | Duration of enrollment = 30 months
  Structured measure viewing Jaspr as appropriate using the Intervention Appropriateness Measure (IAM), Likert type scale, higher scores = stronger patient ratings of appropriateness
Feasibility of Jaspr in ED | Duration of enrollment = 30 months
  Structured clinician measure; qualitative review of barriers to implementation using Feasibility of Intervention Measure (FIM)
Usability, clinician | Duration of enrollment = 30 months
  Structured measure of clinicians' perception of the usability of Jaspr using the System Usability Scale (SUS) , Likert type scale, higher scores = stronger clinician ratings of usability
Usability, patient | Duration of enrollment = 30 months
  Structured measure of clinicians' perception of the usability of Jaspr using the System Usability Scale (SUS), Likert type scale, higher scores = stronger patient ratings of usability
System workflow impact, admissions to psychiatric units | During index ED visit= Day 1
  Of patients who meet eligibility criteria for Jaspr, how many (what percentage) get admitted to a psychiatric unit from the index ED visit, binary, psychiatric hospitalization = yes/No
System workflow impact, door to behavioral health evaluation | During index ED visit= Day 1
  Of patients who meet eligibility criteria for Jaspr, how long in minutes does it take to get a behavioral health evaluation from when they are registered in the ED, continuous, measured in minutes, higher minutes = longer evaluation wait
System workflow impact, total length of stay | During index ED visit= Day 1
  Of patients who meet eligibility criteria for Jaspr, how long in minutes does it take for their entire visit from registration to discharge, continuous, measured in minutes, higher minutes = longer total length of stay
System workflow impact, 28 day revisit | Within 28 days of index ED visit
  Of patients who meet eligibility criteria for Jaspr, how many return to the ED within 28 days, binary, Yes/No
System workflow impact, clinician perception | Assessed within 3 months of Jaspr implementation
  Clinician perception of workflow impact after Jaspr is implemented, assessed by a structured interview, qualitative descriptions

CONTACTS AND LOCATIONS:
Overall Officials: Edwin D Boudreaux, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- UMass Memorial Health, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will comply with the expectations of the NIMH Data Archive (NDA) regarding data components and support documents, including the recommended timeline
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Based on NIMH NDA expectations, investigators will begin sharing data and share data with as long as is expected by NIMH
Access Criteria: See NDA application for details.
URL: https://nda.nih.gov/edit_collection.html?id=4744

REFERENCES:
- See also: The Center for Accelerating Practices to End Suicide through Technology Translation (CAPES)- Signature Project — https://reporter.nih.gov/search/ghz0ZwiyvU2Qfb-N0aHjxw/project-details/10577120